CLINICAL TRIAL: NCT02344069
Title: Effect of Immediate, Pre-emptive Fibrinogen Concentrate in Patients With Trauma Haemorrhage Needing Haemostatic Resuscitation - a Randomized, Controlled, Double-blinded Investigator-initiated Pilot Trial
Brief Title: Pilot Randomized Trial of Fibrinogen in Trauma Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Jakob Stensballe, MD, PhD, Consultant Anaesthetist, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRooF-iTH; 2014-003978-16 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-01-22 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Trauma; Haemorrhage
Keywords: Fibrinogen
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage | interventions — Fibrinogen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrinogen (Active Comparator): Immediate intravenous administration as a single dose of fibrinogen concentrate (Riastap®, CSL Behring), when haemostatic resuscitation is deemed necessary by the clinician.
  Interventions: Drug: Fibrinogen
- Placebo (Placebo Comparator): Saline 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fibrinogen — Human fibrinogen concentrate as a injection
  Other Names: Riastap®, CSL Behring
  Arms: Fibrinogen
Drug: Placebo — Saline 0.9% as a injection
  Other Names: Saline 0.9%
  Arms: Placebo

SUMMARY:
Effect of immediate, pre-emptive fibrinogen concentrate in patients with trauma haemorrhage needing haemostatic resuscitation - a randomized, controlled, double-blinded investigator-initiated pilot trial

DETAILED DESCRIPTION:
Objective To assess the efficacy and safety of an immediate pre-emptive first-line treatment with fibrinogen concentrate in patients with trauma haemorrhage in need of haemostatic resuscitation.

Hypothesis Immediate, pre-emptive first-line treatment of fibrinogen concentrate in trauma patients with ongoing critical haemorrhage will increase the clot strength.

Background Trauma haemorrhage remains a leading cause of morbidity and mortality. Fibrinogen is an essential endogenous component of haemostasis and the plasma level is associated to bleeding, transfusion and outcome.

Trial rationale Fibrinogen concentrate is widely used to correct acquired hypofibrinogenaemia, recommended by several international guidelines including in trauma, but evidence is lacking regarding the treatment safety and efficacy.

Trial population The trial population are patients' ≥ 18 years admitted to the Trauma Centre at Rigshospitalet with immediate need for blood transfusion at arrival and an expected need for haemostatic resuscitation with multiple transfusions during the initial resuscitation. Estimated 30-day mortality is 20 % in the population. Patients included in the trial will be temporarily incompetent because of acute, severe illness related to the ongoing critical bleeding needing multiple transfusion and immediate intervention to control bleeding.

Trial design This is a single centre, randomized (1:1, active:placebo), placebo controlled, double-blind investigator-initiated phase II trial in patients with traumatic, critical bleeding, investigating the safety and efficacy of immediate and pre-emptive administration of fibrinogen concentrate (Riastap®) or placebo as i.v infusion in 40 patients. All patients will receive standard of care including damage control surgery, radiological interventions and haemostatic resuscitation as part of their treatment at Rigshospitalet.

Patients considered to be included in the trial will be temporarily incompetent because of the acute, critical bleeding related to trauma, so scientific guardians will co-sign the informed consent form. Next-of-kin and the patients' general practitioner or the patients will co-sign as soon as possible.

During the study blood samples will be taken at different time points. Patients will be observed and assessed continuously throughout the first 72 hours. During the extended follow up period at day 30, contact will be made with the patients to follow up on safety events and establish potential mortality.

Investigational product Immediate intravenous administration as a single dose of fibrinogen concentrate (Riastap®, CSL Behring), when haemostatic resuscitation is deemed necessary by the clinician. The aim is to give the intervention < 1 hour of arrival, and the intervention should, when possible, be given prior to blood products.

Placebo and blinding Saline 0.9% will be used as placebo. The volume of placebo to be administered is equal to the volume active drug administered. The content (Riastap® or placebo) will be provided in opaque syringes and infusion sets (yellow-coloured) to disguise the content of the allocation to the treatment team.

Outcome measures

Primary outcome measure:

• Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm at 15 min post intervention

Secondary outcome measures:

* TEG® FF MA in mm at 2, 6, 24 and 72 hours post intervention
* TEG® MA in mm at 15 min., 2, 6, 24 and 72 hours post intervention
* Transfusion requirements (Red blood cells (RBC) or fresh frozen plasma (FFP) or platelets (PLT)) at 2, 6, 24, 72 hours and in total at day 30
* Total use of haemostatic therapy (i.e. use of coagulation factor concentrates and tranexamic acid) in the first 24 and 72 hours, omitted from this is active treatment (intervention)
* Time to intervention or placebo
* Time to FFP and PLT transfusion
* Percentage of patients receiving intervention or placebo < 1 hour of arrival
* Time to surgical control of bleeding as noted by the surgeon
* Severe adverse reactions at day 30, defined as symptomatic thromboembolism at day 30 and anaphylaxis at day 30
* 24-hour and 30-day mortality

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient received directly from the scene of the accident AND
* Age ≥ 18 years AND
* Initiated order of transfusion of at least one blood component within the 1st hour of arrival AND
* Predicted to need transfusion package therapy during the initial resuscitation (first 2 hours) AND
* Consent obtainable from patient or scientific guardians (independent physicians and/or next of kin

Exclusion Criteria:

* Duration of > 2 hours from time of accident to arrival at trauma centre OR
* Known anticoagulant treatment (vitamin K antagonist, dabigatran, rivaroxiban, apixaban) OR
* Severe isolated traumatic brain injury OR
* Moribund patient with devastating injuries and expected to die within one hour of admission OR
* Withdrawal from active therapy OR
* Previously, within 30 days, included in a randomized trial, if known at the time of enrolment OR
* Known body weight < 55 kg OR
* Any blood product prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
TEG® Functional Fibrinogen maximum amplitude 15 min | 15 min after intervention
  Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm

SECONDARY OUTCOMES:
TEG® Functional Fibrinogen maximum amplitude 2 hours | 2 hours after intervention
  Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm
TEG® Functional Fibrinogen maximum amplitude 6 hours | 6 hours after intervention
  Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm
TEG® Functional Fibrinogen maximum amplitude 24 hours | 24 hours after intervention
  Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm
TEG® Functional Fibrinogen maximum amplitude 72 hours | 72 hours after intervention
  Thrombelastograph (TEG®) Functional Fibrinogen (FF) maximum amplitude (MA) in mm
TEG® maximum amplitude 15 min | 15 min after intervention
  Thrombelastograph (TEG®) maximum amplitude (MA) in mm
TEG® maximum amplitude 2 hours | 2 hours after intervention
  Thrombelastograph (TEG®) maximum amplitude (MA) in mm
TEG® maximum amplitude 6 hours | 6 hours after intervention
  Thrombelastograph (TEG®) maximum amplitude (MA) in mm
TEG® maximum amplitude 24 hours | 24 hours after intervention
  Thrombelastograph (TEG®) maximum amplitude (MA) in mm
TEG® maximum amplitude 72 hours | 72 hours after intervention
  Thrombelastograph (TEG®) maximum amplitude (MA) in mm
Transfusions requirements | 2, 6, 24, 72 hours and in total at day 30
  Transfusion requirements (Red blood cells (RBC) or fresh frozen plasma (FFP) or platelets (PLT)) at 2, 6, 24, 72 hours and in total at day 30
Total use of haemostatic therapy | 24 hours and 27 hours
  Total use of haemostatic therapy (i.e. use of coagulation factor concentrates and tranexamic acid) in the first 24 and 72 hours, omitted from this is active treatment (intervention)
Time to intervention or placebo | No of minutes from arrival, an expected average of 45 minutes
  Time from arrival to active intervention or placebo in minutes
Time to FFP and PLT transfusion | No of minutes from arrival, an expected average of 50 minutes
  Time to FFP and PLT transfusion in minutes
Percentage of patients receiving intervention or placebo < 1 hour of arrival | 60 min from arrival
  Percentage of patients receiving intervention or placebo < 1 hour of arrival
Time to surgical control of bleeding | No of minutes from arrival, an expected average of 120 minutes
  Time to surgical control of bleeding as noted by the surgeon
Thromboembolism day 30 | 30 days
  Symptomatic thromboembolism at day 30 (Severe adverse reaction)
Anaphylaxis day 30 | 30 days
  Anaphylaxis day 30 (Severe adverse reaction)
24-hour mortality | 24 hours from arrival
  Mortality in the first 24 hours
30-day mortality | 30 days from arrival
  Mortality in the first 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stensballe, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steinmetz J, Sorensen AM, Henriksen HH, Lange T, Larsen CF, Johansson PI, Stensballe J. Pilot Randomized trial of Fibrinogen in Trauma Haemorrhage (PRooF-iTH): study protocol for a randomized controlled trial. Trials. 2016 Jul 19;17(1):327. doi: 10.1186/s13063-016-1439-5. PMID 27430210